CLINICAL TRIAL: NCT06644638
Title: Real-World Persistence and Adherence of Ofatumumab Compared to Self-Injectable and Oral DMTs in Patients With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: COMB157GUS31
Record Dates: First submitted 2024-10-15; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Ofatumumab and Self-injectable DMT Cohort: Adult patients with multiple sclerosis (MS) who newly initiated ofatumumab or other self-injectable DMTs.
- Ofatumumab and Oral DMT Cohort: Adult patients with MS who newly initiated OMB or oral DMTs.

SUMMARY:
This was a retrospective cohort study utilizing the IQVIA PharMetrics® Plus claims database from 01 August 2019 through 31 May 2022.

The database is comprised of fully adjudicated (i.e., paid by the health plan) medical and pharmacy claims and is representative of the commercially insured United States population. Adults treated with ofatumumab (OMB), oral disease-modifying therapies (DMTs) (dimethyl fumarate, diroximel fumarate, monomethyl fumarate, fingolimod, siponimod, ozanimod, ponesimod, teriflunomide, cladribine) or platform self-injectable DMTs (glatiramer acetate, interferon beta-1a, peginterferon beta-1a, interferon beta-1b) between 01 August 2020, through 30 November 2021, were identified. The date of the first incident DMT (OMB, oral DMT, or injectable DMT) during the identification window served as the index date. The baseline period was the 12 months before the index date, and the follow-up period was at least 6 months after the index date. Patients treated with OMB were selected first to maximize sample size, and these patients were allowed to have an oral or injectable DMT in the baseline period. Patients without OMB use during the identification period were categorized into the oral DMT or platform self-injectable DMT cohort based on the first-observed incident DMT during the identification period. For the purpose of this study, platform self-injectable DMTs were referred to as 'self-injectable DMTs.'

ELIGIBILITY:
Inclusion criteria:

* Patients with 1 claim or more for ofatumumab, a newly initiated oral DMT (dimethyl fumarate, fingolimod, teriflunomide, cladribine, siponimod, ozanimod, diroximel fumarate, monomethyl fumarate, ponesimod) or a newly initiated self-injectable DMT (daclizumab, glatiramer acetate, interferon beta-1a, peginterferon beta-1a, interferon beta-1b) occurring during the index window.
* Patients with 12 months or more of pre-index continuous enrollment [CE] with medical and pharmacy benefits.
* Patients with 6 months or more of post-index CE with medical and pharmacy benefits.
* Patients with 2 or more non-ancillary outpatient medical claims (at least 30 days apart) with a diagnosis code for MS (International Classification of Diseases, 10th Revision, Clinical Modification [ICD-10-CM] code: G35) in any position or 1 or more inpatient claims with a diagnosis of MS in the first position during pre-index period.
* No data quality issues (defined as missing age or sex).
* Having two DMTs on the same day was very rare in MS patients per clinician's inputs, but if it happened, those patients were excluded from analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 3632 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Number of Patients Persistent on Ofatumumab and Self-injectable Disease-modifying Therapies (DMTs) | Month 6, month 12
  Persistence was defined as no evidence of discontinuation of the therapy over the follow-up period. Self-injectable DMTs included daclizumab, glatiramer acetate, interferon beta-1a, peginterferon beta-1a, and interferon beta-1b.

OTHER OUTCOMES:
Number of Patients Persistent on Ofatumumab and Oral Disease-Modifying Therapies (DMTs) | Month 6, month 12
  Persistence was defined as no evidence of discontinuation of the therapy over the follow-up period. Oral DMTs included dimethyl fumarate, diroximel fumarate, monomethyl fumarate, fingolimod, siponimod, ozanimod, ponesimod, teriflunomide, and cladribine.
Number of Patients Adherent on Ofatumumab and Oral DMTs | Month 6, month 12
  Adherence was based on the proportion of days covered (PDC), calculated as the number of days with the drug on hand divided by the total number of days in the follow-up period. Oral DMTs included dimethyl fumarate, diroximel fumarate, monomethyl fumarate, fingolimod, siponimod, ozanimod, ponesimod, teriflunomide, and cladribine.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States